CLINICAL TRIAL: NCT03031340
Title: Double Blinded, Randomized, Placebo Controlled Study in Evaluating the Role of Pregabalin in Reducing Opioid Requirement in Spinal Fusion Surgeries of Two or More Vertebrae
Brief Title: Evaluating the Role of Pregabalin in Reducing Opioid Requirement in Spinal Fusion Surgeries of Two or More Vertebrae
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Incidence of AE
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Singh Nair, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-01-004
Record Dates: First submitted 2017-01-22; First posted 2017-01-25 (Estimated); Results first posted 2018-10-10 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Spinal Fusion
Keywords: Spinal fusion; pregabalin; Spinal fusion surgeries; two or more vertebrae
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: placebo
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Pregabalin — On the day of the surgery, 1hour + 15 minutes before the surgery starts, the subject will receive either 300mg of pregabalin or a similarly packaged placebo. On post operative day one, 150 mg of pregabalin or placebo will be given in two doses 12hrs apart.
  Arms: Pregabalin
Other: placebo — placebo
  Arms: Placebo

SUMMARY:
To see if the administration of 3 dosses of pregabalin (1 dose preoperative, 2 doses postoperative) will reduce the postoperative opiate requirements of patients undergoing spinal fusion surgeries of two or more vertebrae.

DETAILED DESCRIPTION:
Introduction

Postoperative pain is often thought to be inadequately treated in half of all surgical procedures . Postoperative pain management in patients undergoing spine surgery is often difficult and challenging. The challenges of opioid tolerance and paucity of efficient opioid sparing agents makes pain management even more complex. Preoperative strategies that can minimize postoperative pain include proper surgical technique, which would avoid or lessen nerve injury, and the use of preemptive analgesia. Studies have shown that the intensity of acute postoperative pain correlates with the risk of developing persistent pain. Post operative pain results from the direct activation of nociceptors, inflammation, and in some cases direct nerve injury to the nerves.

The data on preemptive analgesia are inconclusive . The concept, however, has sparked interest in mechanism-based analgesia and highlighted the process of central sensitization as a target for analgesic intervention .

The use of opioids is limited by their side effect profile and by the poor response of certain types of pain . The multiplicity of mechanisms involved in pain suggests that combination of opioid and non-opioid analgesic drugs will enhance analgesia. The concomitant reduction in opioid requirements, anticipated with the use of multimodal therapy, can also be expected to reduce side effects.

Pregabalin is a lipophilic gamma-amino-butyric acid (GABA) analog with anticonvulsant, anxiolytic and sleep-modulating properties. The effectiveness of pregabalin has been demonstrated in several pain models including neuropathic pain , , incisional injury and inflammation . Several previous studies conducted found that the use of gabapentin, the predecessor of pregabalin, reduced post operative pain and opioid requirements and decreased the number of opioid related adverse events , . Pregabalin is the pharmacologically active S enantiomer of 3-aminomethyl-5-methyl hexanoic acid; it has a similar pharmacological profile to gabapentin . Like gabapentin, pregabalin also binds to the α-2-δ subunit of voltage gated calcium channels, reducing the release of excitatory neurotransmitters: glutamate, norepinephrine, serotonin, dopamine and substance-P. It blocks the development of hyperalgesia and inhibits central sensitization , . Pregabalin has greater absorption, bioavailability, anticonvulsant, anti-hyperalgesic and anxiolytic properties than gabapentin , .

Rationale for selecting spine surgeries. Low back pain is a major medical problem and a significant source of disability for people under 45 years of age . Spine surgeries are considered to be among the most complex, and long-lasting. The postoperative period is particularly challenging for efficient pain management. Postoperative pain may be due to nociceptive pain as well as hyperalgesia secondary to surgical trauma. Central sensitization is a key mechanism in the development and maintenance of chronic pain, particularly for neuropathic pain and pain after spine surgery .

Rationale for using pregabalin

Animal studies in surgical pain models and clinical studies of inflammatory pain in volunteers demonstrated that both of these interventions can cause allodynia and hyperalgesia- these are both susceptible to pregabalin and its analogues , .

The sensitization of dorsal horn neurons has been demonstrated in acute pain models and may be responsible for the development of chronic pain after surgery , , . The ability of pregabalin to reduce the hyperexcitability of dorsal neurons induced by tissue damage confirms its role in preemptive analgesia . Its anxiolytic effect and ability to prevent opioid tolerance could also be beneficial . Alternately, antihyperalgesia drugs like pregabalin may block pathological pain, while leaving the physiological pain (with its protective function) intact. This class of agents function through opiate independent pathways and do not affect gut motility .

Pharmacodynamics and Pharmacokinetics:

Pregabalin is an FDA-approved drug available in 50-300 mg/day (the FDA-recommended maximum is 300mg/day). It is rapidly absorbed following oral administration with peak plasma concentration occurring between 0.7-1.3hrs. The mean oral bioavailability is 90% after 1-300mg of single oral dose. The elimination half-life is 5.5-6.5 hrs independent of dose and repeated administration. Plasma clearance is essentially equivalent to renal clearance. The elimination rate is nearly proportional to creatinine clearance and dose reduction is recommended in patients with low creatinine clearance. Ninety percent of the dose is excreted in the urine .

Adverse events of pregabalin Pregabalin is generally well tolerated and associated with mild to moderate adverse events which are dose dependent. The most frequently reported (22-29%) are dizziness and somnolence. Other less common adverse events reported are dry mouth, peripheral edema, blurred vision and inability to concentrate .

Hypothesis:

Our hypothesis is that pre-operative administration of pregabalin can reduce the central neural sensitization, efficiently reverse inflammatory hyperalgesia and can cause opioid sparing effect. These actions of pregabalin will reduce the amount of opioids need by the patient intraoperatively and in the immediate postoperative period. The reduction of opioids will lessen opioid related adverse events and will augment the perioperative satisfaction level.

ELIGIBILITY:
Inclusion Criteria:

* Age : > 18 years old
* Fusion of > two vertebrae
* Capacity to provide consent
* ASA I-IV
* Ability to swallow capsules

Exclusion Criteria:

* Plan of care includes intubated ICU admission post-op
* Allergy to gabapentin or pregabalin
* Two week prior use of pregabalin
* Significant renal dysfunction (creatinine level >2)
* Severe cardiovascular disease
* History of frequent headaches or dizziness
* Significant hepatic dysfunction (LFT's > 4 times the normal ranges)
* Active usage of alcohol or illicit substances three days prior to surgery
* History of seizure disorders
* Taking medication for anxiety, antiseizure, and psychiatric diagnoses
* Re-operation patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Pregabalin
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Pregabalin | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Opioid Requirement
Description: The primary objective of this study is to evaluate the role of three doses of pregabalin on intra and postoperative (48hrs) opioid requirements in patients undergoing fusion of two or more vertebrae.
Time Frame: 48 hours
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pain Using the Visual Analog Scale (VAS) Pain Score
Description: evaluate pain using the visual analog scale (VAS) pain score at two hrs post-op, the morning following surgery 24 hours and 48 hours post-op
Time Frame: 2 hours, 24 hours, 48 hours
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of 48 Hours Post Operative Nausea and Vomiting
Description: Find the incidence of 48 hours post operative nausea and vomiting in the target population
Time Frame: 48 hours
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Post Operative Cognitive Function
Description: 48 hours post operative headache, dizziness, sedation and blurred vision
Time Frame: 48 hours
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Pre-operative Anxiety
Description: Measure the level of pre-operative anxiety using the visual analog scale (VAS)
Time Frame: 24 hours prior to surgery
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Anesthesia Satisfaction
Description: To measure the level of overall anesthesia satisfaction among the two groups at discharge.
Time Frame: 24 hours post surgery
Population: Data not collected therefore no analysis
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo | Pregabalin
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | Pregabalin (N=1)
Death (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes